CLINICAL TRIAL: NCT07204210
Title: Comparison of Treatment Efficacy of Extracorporeal Shockwave Therapy (ESWT) and Myofascial Release Techniques in Patients With Plantar Fasciitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Burak YİGİT, principal investigator, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRU-FTR-BY-01
Record Dates: First submitted 2025-09-17; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Plantar Fasciitis
Keywords: plantar fascitis; heel pain; myofascial release; eswt; heel spur
MeSH Terms: conditions — Fasciitis, Plantar; Heel Spur | interventions — Extracorporeal Shockwave Therapy; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT treatment group (Experimental): Patients in the ESWT group will receive a total of five sessions of ESWT, once a week for five weeks. The ESWT group will receive 2000 pulses per session at 14 Hz, 2.0 barr intensity, and a dose of 0.2 mJ/mm2. ESWT will be applied primarily to areas near the calcaneal insertion of the plantar fascia.
  Interventions: Device: extracorporeal shockwave therapy
- myofascial release treatment group (Experimental): Myofascial Release treatment group patients will receive treatments once a week for 5 weeks, for a total of 5 weeks. Treatments will be applied once a week for 5 weeks. The following will be applied for a total of 16 minutes: 2 minutes of constant pressure with the therapist's two thumbs to the center of the central part of the plantar fascia and the calcaneal insertion point; 2 minutes of constant pressure with the therapist's thumb to the lateral and medial parts of the plantar fascia, along the line, progressing anteriorly as the fascial tissue relaxes; 2 minutes of constant pressure with the therapist's thumb to the gastrocnemius muscle at its most swollen or taut point, progressing from caudal to cranial with constant pressure from the caudal to cranial point as the tissue relaxes; 2 minutes of constant pressure with the therapist's fist to the central tendon of the plantar fascia; and 2 minutes of constant pressure with the therapist's fist to the gastrocnemius muscle, from caud
  Interventions: Other: myofascial release technique
- control group (Placebo Comparator): Control group patients will not receive any treatment. After the data used in the study is collected, an appointment will be scheduled for five weeks later for comparison. Data will be collected and recorded again after five weeks.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Device: extracorporeal shockwave therapy — Extracorporeal shockwave therapy (ESWT) is a treatment using powerful acoustic pulses which is mostly used to treat kidney stones and in physical therapy and orthopedics. Extracorporeal shockwave therapy is used as a second line measure to treat tennis elbow, shoulder rotator cuff pain, Achilles tendinitis, plantar fasciitis, and greater trochanteric pain syndrome. The lithotripter attempts to break up the stone with minimal collateral damage by using an externally applied, focused, high-intensity acoustic pulse. The patient is usually sedated or anesthetized for the procedure in order to help them remain still and reduce possible discomfort.
  Arms: ESWT treatment group
Other: myofascial release technique — Myofascial release (MFR, self-myofascial release) is an alternative medicine therapy claimed to be useful for treating skeletal muscle immobility and pain by relaxing contracted muscles, improving blood and lymphatic circulation and stimulating the stretch reflex in muscles. Writing for Science-Based Medicine, Harriet Hall described myofascial release as an umbrella term for several types of physical manipulation, which might more simply be described as a kind of massage based on vaguely defined scientific notions. Reviews published in 2013 and 2015 evaluating evidence for MFR efficacy found that clinical trials that had been conducted varied in quality, technique, outcome measurements and had mixed outcomes; the 2015 review noted: "it is time for scientific evidences on MFR to support its clinical use.
  Arms: myofascial release treatment group
Other: Placebo Control — Participants were not given any interventions that had proven effective for treatment. An appointment was made for 5 weeks later.
  Arms: control group

SUMMARY:
Various treatment methods are employed for patients diagnosed with plantar fasciitis. However, many of these approaches involve high-cost interventions, such as extracorporeal shock wave therapy (ESWT) and platelet-rich plasma (PRP) applications. The present study aims to compare the treatment effectiveness of myofascial release-considered a cost-effective intervention-with ESWT, which is among the most commonly preferred treatment modalities.

DETAILED DESCRIPTION:
The present study aims to compare the effectiveness of extracorporeal shock wave therapy (ESWT), a frequently used treatment for patients with plantar fasciitis and heel pain, with specific myofascial release techniques. The paucity of studies in the literature and the lack of definitive evidence on this topic served as the basis for initiating this research. A total of 114 patients diagnosed with plantar fasciitis, deemed appropriate for ESWT and myofascial release therapy and meeting the inclusion criteria, are planned to participate in the study. These 114 patients will be randomly divided into three groups of 38 each. Before and after treatment, each patient will complete a demographic data form, the Visual Analog Scale (VAS), the Foot Function Index (FFI), the Roles and Maudsley pain scores, and the American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot clinical assessment scales. Participants will be randomly selected from among individuals who applied to Kayseri City Hospital with complaints of plantar fasciitis within the Kayseri province. The three groups will consist of a myofascial release treatment group, an ESWT treatment group, and a control group. The ESWT group will receive 2,000 pulses per session at 2.0 bar intensity, 14 Hz frequency, and a dose of 0.2 mJ/mm². Specific myofascial release techniques will be administered to the myofascial release group once per week for 16 minutes, over a total period of 5 weeks. No treatment will be administered to the control group. An evaluation appointment will be scheduled 5 weeks after baseline data collection using the designated assessment tools. Pre-treatment and post-treatment data for all three groups will be recorded using the SPSS software. After data collection is completed, appropriate statistical analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being able to communicate in Turkish
* Being able to read and write
* Voluntarily agreeing to participate in the study
* Having been diagnosed with plantar fasciitis

Exclusion Criteria:

* Obvious major foot trauma
* Pregnancy
* Presence of tumor
* Coagulation disorder
* Presence of open wounds and extreme sensitivity in the foot area
* Having had any surgical operation on the foot and ankle
* Partial amputation of the foot
* Application of one and/or more physical medicine modalities and corticosteroid injections within the last 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-27 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society Ankle-Hindfoot Scale (AOFAS-AHFS) | pre-treatment, 1st week post-treatment and 6th week post-treatment
  The AOFAS-hindfoot clinical assessment system grades the ankle, subtalar, talonavicular, and calcaneocuboid joint levels. A patient can receive a score of 100 if they have no pain, full sagittal and hindfoot range of motion, no instability in the ankle or hindfoot, good alignment, the ability to walk more than six blocks, the ability to walk on any walking surface, no noticeable limp, no limitations in daily or recreational activities, and no need for assistive devices for ambulation. The scale includes 50 points for function, 40 points for pain, and 10 points for alignment. Increasing scores indicate that the patient's condition is good.
Foot Function İndex (FFİ) | pre-treatment, 1st week post-treatment and 6th week post-treatment
  447 / 5.000 The Foot Function Index (FFI) is a questionnaire that assesses multiple dimensions of foot function. The FFI consists of 23 items divided into three subscales that measure the impact of foot pathology on pain, disability, and activity limitation. The Foot Function Index is widely used in various pathologies and treatments related to foot and ankle problems, including congenital, acute, and chronic diseases, injuries, and surgical procedures. Increasing scores indicate that the patient's condition is good.
Visual Analog Scale (VAS) | pre-treatment, 1st week post-treatment and 6th week post-treatment
  This scale was created to assess the severity of pain in patients. Patients will be asked to rate their heel and sole pain on a scale of 1 to 10. 10 represents severe, function-limiting, and unbearable pain, while 0 represents no pain at all.

SECONDARY OUTCOMES:
Roles and Maudsley pain score | pre-treatment, 1st week post-treatment and 6th week post-treatment
  The Roles and Maudsley pain scoring is a method used to assess pain level and range of motion. This score is divided into four categories:
  Excellent (1 Point): No pain, full range of motion, and activity. Good (2 Points): Occasional discomfort, full range of motion, and activity. Fair (3 Points): Some pain after prolonged activity. Poor (4 Points): Pain that limits activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No